CLINICAL TRIAL: NCT02999958
Title: Comparison of G-Series Media System With Antioxidants Versus Standard G-Series Media System
Brief Title: Adding Antioxidants Into Human Sequential Culture Media System
Acronym: Antioxidants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitrolife (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AOX-G_Series-2016
Record Dates: First submitted 2016-12-16; First posted 2016-12-21 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Culture Media; Blastocyst; Antioxidants; Embryo; Human; Oxygen
MeSH Terms: interventions — Antioxidants; Acetylcarnitine; Acetylcysteine; Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Sequential culture media without addition of antioxidants
- Treatment (Active Comparator): Sequential culture media with the addition of antioxidants
  Interventions: Biological: Antioxidants

INTERVENTIONS:
Biological: Antioxidants — In the Treatment Arm, the G-Series culture media system will be used with antioxidants
  Other Names: Acetyl-L-carnitine (ALC); N-acetyl-L-cysteine (NAC); alpha-Lipoic acid (ALA)
  Arms: Treatment

SUMMARY:
Upon collection, human oocytes are fertilized and culture up to the blastocyst stage, followed by transfer and / or cryopreservation. Culture media systems have been developed that support each step of this process. Although these culture media systems try to mimic the natural environment, several components of the in-vivo situation are not present in today´s media. One such component is anti-oxidants that may protect embryos against damage by reactive oxygen species.

This investigation aims to compare blastocyst development using 2 different types of culture media systems, one of which contains antioxidants. Patients having at least eight oocytes and meeting other inclusion criteria can be included in this investigation.

It is a prospective randomized multicenter study randomly dividing oocytes into two groups and assessing parameters of embryo development from fertilization up to blastocyst formation until day six. Embryos with acceptable developmental characteristics can be transferred into the uterus or cryopreserved for later use.

The investigation is designed as a superiority study comparing utilization rate of blastocysts per normally fertilized oocyte using both media systems. In patients receiving embryo transfer in the fresh treatment cycle, detection of clinical pregnancy by ultrasound after 12 weeks gestation is the final endpoint of the investigation.

DETAILED DESCRIPTION:
Study objective:

Study comparing blastocyst development on the same cohort of oocytes using two different media systems, sequential G-Series media versus sequential G-Series media supplemented with antioxidants.

Primary endpoint:

Percentage of good quality blastocysts (GQB) per fertilized oocyte on day 5.

Secondary endpoints:

Embryo development day 3, 5 and 6 Embryo quality day 3, 5 and 6 Total blastocyst formation (day 5 and day 6) Utilization rate (embryos available for transfer and cryopreservation) Biochemical pregnancy rate Implantation rate Clinical pregnancy rate

Setup:

Prospective oocyte sibling, superiority study

MATERIALS AND METHODS

Intervention:

New type of embryo culture media used for in vitro culture of human IVF embryos.

Power analysis:

The planning and the power analysis was made together with a statistician, Nils-Gunnar Pehrsson.

From retrospective data using simulation, the intra individual SD for the difference in % GQB between the two media strategies was estimated to 32%. In order to find a difference in 8% in GQB between the two media with power 80% with paired T-test 128 couples will be needed.

Randomization:

Couples will be enrolled in the study at oocyte pick up (day 0). A minimum of 8 cumulus-oocyte-complexes is required for participation.

Stratified randomization of the oocytes by couple will be performed. For each couple the oocytes will be numbered.

These oocytes for each couple will then be block (by two) randomized to the two media types; A (Traditional G-Series media system = Control) and B (G-Series media system with antioxidant = intervention). In both groups traditional culture will be performed. Allocation will be performed in a 1:1 ratio according to a unique randomization list for each couple.

Blinding:

To minimize possible bias for the primary outcome (GQB D5) the embryologist performing the morphological evaluation on day 5/6 will not know which group the embryos belong to.

Both the physician and the couple will be blinded in respect to from which group an embryo was selected for transfer.

IVF treatment procedure:

A traditional IVF treatment will be performed including ovarian stimulation and oocyte pick-up using the standard methods at the clinics.

Embryo assessment on day 3 according to Alpha/ESHRE consensus criteria and on day 5 according to Gardner score.

Morphological scoring Embryo development and morphology on day 3 will be scored based on the Alpha/ESHRE Consensus criteria. Blastocyst development and morphology will be scored according to a published scoring system for blastocysts and will be documented with individual photos of each blastocyst. Embryo & Blastocyst scoring will be performed under an inverted microscope on day 3 and days 5 & 6, respectively. Blastocysts that have a score equal or higher than 3BB are considered as GQB.

DOCUMENTATION All patients participating in the study will be documented on a computerized CRF. This document will contain study-specific relevant clinical and laboratory data from the specific IVF cycle.

STATISTICAL ANALYSIS Both an Intention-to-Treat (ITT) population and a Per Protocol (PP) population will be defined. Primary efficacy variable in this superiority study will be difference in % GQB between the two media types for each couple. Primary statistical analysis will be two-sided paired T-test regarding the mean of difference in % GQB between Standard sequential culture media and Antioxidant media on the ITT population. A two sided 95% confidence interval for the mean difference in % GOB between the two media will be calculated. All significance tests will be two-sided and conducted at the 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* Minimum eight cumulus-oocyte-complexes.
* Couples with female, male or unexplained infertility intending to undergo IVF
* The couple should have received verbal and written information/consent about the study.
* Blastocyst culture and embryo transfer is decided.
* If the couple fulfills the criteria above their consent to participate must be given and documented in the couple's medical journal.

Exclusion Criteria:

* Previous participation in the study
* PGD/PGS
* Surgically retrieved sperm cells (TESA / TESE)
* If split IVF is needed
* Less than eight cumulus-oocyte-complexes
* More than thirty cumulus-oocyte-complexes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Percentage of good quality blastocyst (GQB) per fertilized oocyte on day 5 | 7 months

SECONDARY OUTCOMES:
Embryo development on day 3, 5 & 6 | 7 months
Embryo quality on day 3, 5 & 6 | 7 months
Total blastocyst rate | 7 months
Blastocyst utilization rate per fertilized oocyte | 7 months
Biochemical pregnancy rate | 8 months
Clinical pregnancy rate | 9 months
Implantation rate | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: A Yoshida, MD, PhD, Principal Investigator — Kiba Park Clinic, Tokyo
Locations (2):
- Japan (2):
  - Kuramoto Women´s Clinic, Fukuoka
  - Kiba Park Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gardner DK, Lane M, Stevens J, Schlenker T, Schoolcraft WB. Blastocyst score affects implantation and pregnancy outcome: towards a single blastocyst transfer. Fertil Steril. 2000 Jun;73(6):1155-8. doi: 10.1016/s0015-0282(00)00518-5. PMID 10856474